CLINICAL TRIAL: NCT04337697
Title: Neonatal Seizure Registry - Developmental Functional EValuation
Acronym: NSR-DEV
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Michigan (Other); Stanford University (Other); Duke University (Other); Boston Children's Hospital (Other); Children's National Research Institute (Other); Massachusetts General Hospital (Other); Children's Hospital of Philadelphia (Other); Children's Hospital Medical Center, Cincinnati (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-28584; 1R01NS111166-01A1 (NIH); R01NS111166 (NIH)
Record Dates: First submitted 2020-03-31; First posted 2020-04-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Seizure; Hypoxic-Ischemic Encephalopathy; Stroke; Intracranial Hemorrhages; Epilepsy; Cerebral Palsy; Intellectual Disability
Keywords: Family impact; Neurodevelopment
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Stroke; Intracranial Hemorrhages; Epilepsy; Cerebral Palsy; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NSR-DEV study is a longitudinal cohort study of around 280 Neonatal Seizure Registry participants that aims to evaluate childhood outcomes after acute symptomatic neonatal seizures, as well as examine risk factors for developmental disabilities and whether these are modified by parent well-being.

DETAILED DESCRIPTION:
Neonatal seizures due to brain injury (acute symptomatic seizures) are associated with high risk of neurodevelopmental disability in infancy. Although prognosis in early childhood is a critical question for parents and providers, outcomes beyond infancy are largely unknown. Further, parents of infants with neonatal seizures are at risk for mental health disorders, which can undermine their ability to care for a child with medical complexity and may contribute to impaired child development.

The NSR-DEV study is a longitudinal cohort study of around 280 Neonatal Seizure Registry participants enrolled at one of nine sites across the USA. Participants will be evaluated using developmental questionnaires and in-person neurodevelopmental testing. Parent well-being will be assessed at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in NSR-II
* Alive at the start of the NSR-DEV study period
* Parent(s) who are English or Spanish literate (with assistance of interpreter)

Exclusion Criteria:

* Neonates who were found to have exclusion criteria after NSR-II enrollment
* Risk for adverse outcome independent of seizures and underlying brain injury (including but not limited to: inborn errors of metabolism, fetal infection, brain malformation)
* Transient cause for seizures (e.g., mild hypoglycemia, hyponatremia, hypocalcemia with normal neuroimaging)
* Neonatal-onset epilepsy syndromes

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Outpatient, family members/caregivers, providers, children/minors, subjects unable to read, speak or understand English
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Full scale IQ (FSIQ) score for each child on the Wechsler Preschool and Primary Scale of Intelligence, 4th Edition (WPPSI-IV) | At age 5.5 years during in-person study visit
  The WPPSI-IV is an in-person assessment administered by a psychologist or psychometrician that will be used to measure neurocognitive ability. Full Scale IQ (FSIQ) will be generated for each participant from the following subtests: Verbal Comprehension Index (VCI), Visual Spatial Index (VSI), Fluid Reasoning Index (FRI), Working Memory Index (WMI), Processing Speed Index (PSI), Receptive Vocabulary and Picture Naming.

SECONDARY OUTCOMES:
Change in scores over time for each child on the Vineland Adaptive Behavior Scales, 3rd Edition | At enrollment study visit and annual visits when the child is age 3, 4, 5.5, 7, and 8
  The Vineland Adaptive Behavior Scales Parent Form measures adaptive behavior and intellectual and developmental function. Adaptive behavior is predictive of functional performance in school and is linked to both cognitive and executive function. Scores for each participant at each timepoint are generated based on parent reports in the following categories: Communication, Daily Living Skills, Socialization, Motor Skills, Adaptive Behavior Composite (ABC). We will look at the change in score over time for each participant during the study period after the Vineland-3 is administered at each timepoint.

OTHER OUTCOMES:
Scores for each child on Behavior Rating Inventory of Executive Function®, Preschool version (BRIEF-P) | At enrollment study visit
  BRIEF-P is a standardized measure of early childhood executive function. Scores are generated based on parent report of a child's function in the Global Executive Composite (GBC) scale.
Scores for each child on Behavior Rating Inventory of Executive Function®, Preschool version (BRIEF-P) | At age 5.5 years during in-person study visit
  BRIEF-P is a standardized measure of early childhood executive function. Scores are generated based on parent report of a child's function in the Global Executive Composite (GBC) scale.
Scores for each child on The Social Responsiveness Scale, 2nd edition (SRS-2) - Parent Form | At enrollment study visit
  SRS-2 (Parent Form) is an online tool to identify social impairment associated with Autism Spectrum Disorders and quantifies Autism Spectrum Disorder severity. Scores are generated based on parent report of child's function in these scales: Social Awareness, Social Cognition, Social Communication, Social Motivation, Restricted Behaviors and Repetitive Behavior. A total score as well as separate scale scores are generated.
Scores for each child on The Social Responsiveness Scale, 2nd edition (SRS-2) - Parent Form | At age 5.5 years during in-person study visit
  SRS-2 (Parent Form) is an online tool to identify social impairment associated with Autism Spectrum Disorders and quantifies Autism Spectrum Disorder severity. Scores are generated based on parent report of child's function in these scales: Social Awareness, Social Cognition, Social Communication, Social Motivation, Restricted Behaviors and Repetitive Behavior. A total score as well as separate scale scores are generated.
Scores for each child on The Social Responsiveness Scale, 2nd edition (SRS-2) - Teacher Form | At age 5.5 years during in-person study visit
  SRS-2 (Teacher Form) is an online tool to identify social impairment associated with Autism Spectrum Disorders and quantifies Autism Spectrum Disorder severity. Scores are generated based on teacher report of child's function in these scales: Social Awareness, Social Cognition, Social Communication, Social Motivation, Restricted Behaviors and Repetitive Behavior. A total score as well as separate scale scores are generated.
Scores for each child on Behavior Assessment System for Children, 3rd edition (BASC-3) - Parent Form | At enrollment study visit
  BASC-3 (Parent Form) is a measure of both adaptive and problem behaviors. Scores are generated based on parent report of a child's behavior in these scales: Externalizing Problems, Internalizing Problems, Adaptive Skills, Hyperactivity, Attention Problems, Atypicality, and Social Skills.
Scores for each child on Behavior Assessment System for Children, 3rd edition (BASC-3) - Parent Form | At age 5.5 years during in-person study visit
  BASC-3 (Parent Form) is a measure of both adaptive and problem behaviors. Scores are generated based on parent report of a child's behavior in these scales: Externalizing Problems, Internalizing Problems, Adaptive Skills, Hyperactivity, Attention Problems, Atypicality, and Social Skills.
Scores for each child on Behavior Assessment System for Children, 3rd edition (BASC-3) - Teacher Form | At age 5.5 years during in-person study visit
  BASC-3 (Teacher Form) is a measure of both adaptive and problem behaviors. Scores are generated based on teacher report of a child's behavior in these scales: Externalizing Problems, Internalizing Problems, Behavior Symptoms Index, Adaptive Skills, School Problems, Hyperactivity, Attention Problems, Atypicality, and Social Skills.
Scores for each child on Child Sensory Profile, 2nd edition - Parent Form | At enrollment study visit
  Child Sensory Profile, 2nd edition (Parent Form) is a standardized instrument to evaluate sensory processing issues, including oversensitivity to sights, sounds, textures, and other sensory input. Scores are generated based on parent report of child's processing in these areas: Seeking/Seeker, Avoiding/Avoider, Sensitivity/Sensor, Registration/Bystander, Auditory Processing, Visual Processing, Touch Processing, Movement Processing, Body Position Processing, and Oral Sensory Processing.
Scores for each child on Child Sensory Profile, 2nd edition - Parent Form | At age 5.5 years during in-person study visit
  Child Sensory Profile, 2nd edition (Parent Form) is a standardized instrument to evaluate sensory processing issues, including oversensitivity to sights, sounds, textures, and other sensory input. Scores are generated based on parent report of child's processing in these areas: Seeking/Seeker, Avoiding/Avoider, Sensitivity/Sensor, Registration/Bystander, Auditory Processing, Visual Processing, Touch Processing, Movement Processing, Body Position Processing, and Oral Sensory Processing.
Scores for each child on Kaufman Test of Educational Achievement, 3rd edition (KTEA-3) | At age 5.5 years during in-person study visit
  KTEA-3 is a standardized instrument that provides in-depth assessment and evaluation of key academic skills. Scores are generated based on child performance in these areas: Spelling, Letter and Word Recognition and Math Computation.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At enrollment study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At (child) age 3 years during annual study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At (child) age 4 years during annual study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At (child) age 5.5 years during in-person study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At (child) age 7 years during annual study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on Hospital Anxiety Depression Scale (HADS) | At (child) age 8 years during annual study visit
  Hospital Anxiety Depression Scale (HADS) is a well-validated, 14-item, measure of symptoms of anxiety and depression. Scores will be generated based on parent/guardian response to the HADS questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At enrollment study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At (child) age 3 years during annual study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At (child) age 4 years during annual study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At (child) age 5.5 years during in-person study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At (child) age 7 years during annual study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on WHO Quality of Life-BREF (WHOQOL-BREF) | At (child) age 8 years during annual study visit
  WHO Quality of Life-BREF (WHOQOL-BREF) assesses four domains of health: physical, psychological, social relationships, and environment. It also includes two general questions on self-perceived QOL and general health. Scores will be generated based on parent/guardian response to the WHOQOL-BREF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At enrollment study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At (child) age 3 years during annual study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At (child) age 4 years during annual study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At (child) age 5.5 years during in-person study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At (child) age 7 years during annual study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact on Family Scale (IOF) | At (child) age 8 years during annual study visit
  The Impact on Family Scale (IOF) measures parent perception of the ill child's impact on the family. The score represents a construct of personal, family and social impact. Scores will be generated based on parent/guardian response to the IOF questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At enrollment study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At (child) age 3 years during annual study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At (child) age 4 years during annual study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At (child) age 5.5 years during in-person study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At (child) age 7 years during annual study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Impact of Events Scale - Revised | At (child) age 8 years during annual study visit
  The Impact of Events Scale - Revised is a validated measure of post-traumatic stress reactions. Scores will be generated based on parent/guardian response to the Impact of Events Scale - Revised questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At enrollment study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At (child) age 3 years during annual study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At (child) age 4 years during annual study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At (child) age 5.5 years during in-person study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At (child) age 7 years during annual study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Scores for each parent/guardian on The Post Traumatic Growth Inventory | At (child) age 8 years during annual study visit
  The Post Traumatic Growth Inventory is a commonly used, validated measure of resilience that has been incorporated into studies of parents of sick neonates and children. Scores will be generated based on parent/guardian response to The Post Traumatic Growth Inventory questionnaire.
Written responses from each parent/guardian on Open Ended Questions | At enrollment study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.
Written responses from each parent/guardian on Open Ended Questions | At (child) age 3 years during annual study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.
Written responses from each parent/guardian on Open Ended Questions | At (child) age 4 years during annual study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.
Written responses from each parent/guardian on Open Ended Questions | At (child) age 5.5 years during in-person study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.
Written responses from each parent/guardian on Open Ended Questions | At (child) age 7 years during annual study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.
Written responses from each parent/guardian on Open Ended Questions | At (child) age 8 years during annual study visit
  The Open Ended Questions ask parents/guardians to explain different aspects of caring for their child and their child's healthcare journey and for any advice they would give to both the healthcare team and other parents of children with similar conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah C. Glass, MDCM, MAS, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
In accordance with study sponsor
Time Frame: In accordance with study sponsor
Access Criteria: In accordance with study sponsor

REFERENCES:
- [Derived] Franck LS, Lemmon ME, Grossbauer L, Pawlowski K, Sturza JS, Wusthoff CJ, Massey SL, Chu CJ, Soul JS, Numis AL, Thomas C, Benedetti GM, Anwar T, Berl MM, Gidley Larson JC, Rogers EE, Chen C, McCulloch CE, Glass HC, Shellhaas RA. Parent and Family Well-Being and Associated Risk Factors as Children with Neonatal Seizures Reach Preschool and School-Age: A Longitudinal Cohort Study. J Pediatr Clin Pract. 2025 May 16;16:200149. doi: 10.1016/j.jpedcp.2025.200149. eCollection 2025 Jun. PMID 40510235